CLINICAL TRIAL: NCT02469857
Title: Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Study of AB103 as Compared to Placebo in Patients With Necrotizing Soft Tissue Infections. ACCUTE (AB103 Clinical Composite Endpoint Study in Necrotizing Soft Tissue Infections)
Brief Title: Phase III Efficacy and Safety Study of AB103 in the Treatment of Patients With Necrotizing Soft Tissue Infections
Acronym: ACCUTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Atox Bio Ltd (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATB-202
Record Dates: First submitted 2015-06-06; First posted 2015-06-12 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Necrotizing Soft Tissue Infections; Necrotizing Fasciitis; Fournier's Gangrene
Keywords: AB103; Necrotizing fasciitis
MeSH Terms: conditions — Fasciitis, Necrotizing; Fournier Gangrene | interventions — AB103; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AB103 0.5 mg/kg (Experimental): AB103 0.5 mg/kg, IV, single dose
  Interventions: Drug: AB103 0.5 mg/kg
- NaCl 0.9% (Placebo Comparator): NaCl 0.9%, IV, single dose
  Interventions: Other: NaCl 0.9%

INTERVENTIONS:
Drug: AB103 0.5 mg/kg
  Other Names: reltecimod
  Arms: AB103 0.5 mg/kg
Other: NaCl 0.9%
  Other Names: Normal saline
  Arms: NaCl 0.9%

SUMMARY:
The purpose of this study is to determine whether AB103 is safe and effective in the treatment of patients with necrotizing soft tissue infections (NSTI) receiving standard of care therapy.

DETAILED DESCRIPTION:
The primary hypothesis of this study is that in addition to standard of care treatment (which includes surgical intervention, antimicrobial therapy and critical care support for organ dysfunction or failure), AB103 will demonstrate a clinically significant treatment benefit over placebo.

This hypothesis will be addressed by measuring the effect of AB103 on a composite of clinical parameters associated with the disease course of patients with NSTI, using a responder analysis. A responding patient must meet all 5 parameters of the composite clinical success end point, while a non-responding patient can fail by not meeting any one of the parameters. These analyses are designed to demonstrate that in addition to being safe, one dose of 0.5 mg/kg of AB103 will:

Improve systemic signs of the infection by improving organ function of patients compared to placebo as measured by:

* Survival at Day 28
* Modified SOFA (mSOFA) score on Day 14 and change from baseline to Day 14 ≥ 3. A Day 14 mSOFA score of ≤1 and a change from baseline (pre-treatment) to Day 14 ≥3 will be required for a patient to achieve the primary composite clinical success endpoint (NICCE)

Improve the local signs of the infection, as measured by:

* Reduced number of debridements, counted to Day 14. No more than 3 debridements to Day 14 will be required for a patient to achieve composite clinical success
* No amputation after the first debridement (amputation on the first debridement is not considered a failure). A patient will be required to have had no amputations done after the first surgical procedure in order to achieve composite clinical success.

  290 patients will be recruited into the study and randomized to receive either 0.5 mg/kg AB103 or placebo in a 1:1 ratio. Randomization will be stratified within center by the diagnosis of Fournier's Gangrene and mSOFA score category (3-4 vs >4) at screening. The study will be conducted with interim analyses for futility at 100 patients and safety monitored by an independent Data Monitoring Board at regular planned intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Surgical confirmation of NSTI by attending surgeon;
2. mSOFA score ≥3 (in any one or combination of the 5 major components of SOFA score with one organ component having a score of at least 2: cardiovascular, respiratory, renal, coagulation, CNS), measured as close as possible to the first debridement;
3. IV drug administration within 6 hours from the clinical diagnosis and the decision at the study site, to have an urgent surgical exploration and debridement (drug should not be administered until surgical confirmation is established);
4. If a woman is of childbearing potential, she must consistently use an acceptable method of contraception from baseline through Day 28;
5. If a male patient's sexual partner is of childbearing potential, the male patient must acknowledge that they will consistently use an acceptable method of contraception (defined above) from baseline through Day 28.
6. Signed and dated informed consent (ICF) as defined by the Institutional Review Board (IRB) and, if applicable, California Bill of Rights. If patient is unable to comprehend or sign the ICF, patient's legally acceptable representative may sign the ICF

Exclusion Criteria:

1. BMI>51;
2. Patient who has been operated at least once for the current NSTI infection and had a curative deep tissue debridement;
3. Patients with overt peripheral vascular disease in the involved area ;
4. Diabetic patients with peripheral vascular disease who present with below the ankle infection;
5. Removed deep vein thrombosis (DVT) in area of NSTI as an exclusion criteria
6. Patient with burn wounds;
7. Current condition of: (a) Inability to maintain a mean arterial pressure > 50 mmHg and/or systolic blood pressure > 70 mmHg for at least 1 hour prior to screening despite the presence of vasopressors and IV fluids or (b) a patient with respiratory failure such that an SaO2 of 80% cannot be achieved or (c) a patient with refractory coagulopathy (INR >5) or thrombocytopenia (platelet count <20,000) that does not partially correct with administration of appropriate factors or blood products;
8. Chronic neurological impairment that leads to a neuro mSOFA component ≥2;
9. Recent cerebrovascular accident in the last 3 months;
10. Patients with cardiac arrest requiring cardiopulmonary resuscitation within the past 30 days;
11. Patient is not expected to survive throughout 28 days of study due to underlying medical condition, such as poorly controlled neoplasm;
12. Patient or patient's family are not committed to aggressive management of the patient's condition;
13. Any concurrent medical condition, which in the opinion of the Investigator, may compromise the safety of the patient or the objectives of the study or the patient will not benefit from treatment such as:

    * Congestive heart failure (CHF){ New York Heart Association (NYHA) class III-IV}
    * Severe chronic pulmonary obstructive disease (COPD)
    * Liver dysfunction {Childs-Pugh class C}
    * Immunosuppression (see Appendix F, Section 15.6 for list of excluded immunosuppressive medications)
    * Neutropenia < 1,000 cells/mm3not due to the underlying infection
    * Idiopathic Thrombocytopenia Purpura
    * Receiving or about to receive chemotherapy or biologic anti-cancer treatment although hormonal manipulation therapies for breast and prostate malignancies are permitted
    * Hematological and lymphatic malignancies in the last 5 years;
14. Known HIV infection with CD4 (cluster of differentiation 4) count < 200 cells/mm3 or < 14% of all lymphocytes;
15. Patients with known chronic kidney disease (documented pre-illness creatinine value(s) ≥2.0) or patients receiving renal replacement therapy for chronic kidney disease;
16. Patients that are treated with continuous hemofiltration (e.g. Continuous Veno-Venous Hemofiltration) for acute kidney dysfunction, not due to NSTI, starting prior to study drug administration;
17. Pregnant or lactating women;
18. Previous enrollment in a clinical trial involving investigational drug or a medical device within 30 days;
19. Previous enrollment in this protocol, ATB-202 or the Phase 2 trial of AB103, ATB-201.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2019-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne M Dankner, MD, Study Director — Atox Bio Ltd; Eileen M Bulger, MD, Principal Investigator — Harborview Injury Prevention and Research Center
Locations (71):
- United States (61):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Maricopa Medical Center, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Los Angeles Biomedical Research Institute at Harbor UCLA Medical Center, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - UCSD Medical Center, San Diego, California
  - UCH-Memorial Health System, Colorado Springs, Colorado
  - University of Colorado Hospital, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - UF Health Shands Hospital, Gainesville, Florida
  - Ryder Trauma Center/Jackson Memorial Hospital, Miami, Florida
  - Emory University at Grady Memorial Hospital, Atlanta, Georgia
  - Augusta University Health, Augusta, Georgia
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Baton Rouge General Hospital, Baton Rouge, Louisiana
  - LSU Health Science Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University-Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Wayne State University-Sinai Grace Hospital, Detroit, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - St Louis University, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Capital Health System, Inc., Trenton, New Jersey
  - Albany Medical Center, Albany, New York
  - Erie County Medical Center-Affliate of SUNYat Buffalo, Buffalo, New York
  - Staten Island University Hospital-Northwell Health, Staten Island, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati Medical Center (UCMC), Cincinnati, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Wright State University & Premier Health Clinical Trials Research Alliance, Dayton, Ohio
  - St Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Legacy Emanuel Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - The Pennsylvania State University and The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Trauma Center at PENN, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center at El Paso, El Paso, Texas
  - John Peter Smith Health Network, Fort Worth, Texas
  - Baylor College of Medicine-Ben Taub Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Medical Center, Temple, Texas
  - Harborview Medical Center, Seattle, Washington
  - Medical College of Wisconsin-Froedtert Hospital, Milwaukee, Wisconsin
- France (10):
  - Hộpital Estaing-CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hộpital Henri Mondor, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Robert Salengro Hopital-CHRU Lille, Lille
  - CHU de Limoges, Limoges
  - Hôpital Edouard Herriot, Lyon
  - CHRU Nancy, Hôpital Central, Nancy
  - CHU de Nimes, Nîmes
  - Hôpital de la Source, CHR Orleans, Orléans
  - CHRU Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bulger EM, May AK, Robinson BRH, Evans DC, Henry S, Green JM, Toschlog E, Sperry JL, Fagenholz P, Martin ND, Dankner WM, Maislin G, Wilfret D, Bernard AC; ACCUTE Study Investigators. A Novel Immune Modulator for Patients With Necrotizing Soft Tissue Infections (NSTI): Results of a Multicenter, Phase 3 Randomized Controlled Trial of Reltecimod (AB 103). Ann Surg. 2020 Sep 1;272(3):469-478. doi: 10.1097/SLA.0000000000004102. PMID 32657946

RESULTS

PARTICIPANT FLOW:
Groups:
- Reltecimod (AB103) 0.5 mg/kg: Reltecimod 0.5 mg/kg, single IV infusion over approximately 10 minutes
- Placebo: NaCl 0.9%, single IV infusion over approximately 10 minutes
Period: Overall Study
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Started (As Treated (Safety) Analysis Set) | 143 | 147
Completed (As Treated (Safety) Analysis Set) | 118 | 115
Not Completed | 25 | 32
Not completed — Death | 24 | 29
Not completed — Discontinuation | 1 | 3

BASELINE CHARACTERISTICS:
Population: This analysis population (As Treated/Safety Analysis Set) included all randomized patients who were exposed to study drug (reltecimod or placebo), with patients analyzed according to the treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo | Total
Number analyzed (Participants) | 143 | 147 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (15.3) | 56.3 (15.0) | 54.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 117
  Male | 85 | 88 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 131 | 133 | 264
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Instead of collecting data in the categories "More than one race" and "Unknown or Not Reported," data were collected in the categories "Other" and "Missing." Counts of participants in these latter 2 categories were summed and included in the category of "Unknown or Not Reported" in this study record.
  Participants
    American Indian or Alaska Native | 3 | 2 | 5
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 23 | 24 | 47
    White | 106 | 110 | 216
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 9 | 10 | 19
Region of Enrollment [Number; unit: participants] — This measure represents the two countries from which patients were enrolled into this study and received study drug (i.e., United States and France).
  participants
    United States | 135 | 138 | 273
    France | 8 | 9 | 17
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.4 (8.3) | 33.7 (8.3) | 32.5 (8.4)
Necrotizing Soft Tissue Infection (NSTI) Diagnosis [Count of Participants; unit: Participants]
  Necrotizing Fasciitis | 96 | 95 | 191
  Fournier's Gangrene | 43 | 40 | 83
  Gas Gangrene/Myonecrosis | 1 | 4 | 5
  Other NSTI | 3 | 8 | 11
Comorbidities [Count of Participants; unit: Participants]
  Diabetes | 64 | 59 | 123
  Cardiovascular Disease | 37 | 28 | 65
  Smoker | 34 | 32 | 66
  Alcohol Abuse | 17 | 13 | 30
Modified Sequential Organ Failure Assessment (mSOFA) Score [Mean (Standard Deviation); unit: score on a scale] — Modified Sequential Organ Failure Assessment (mSOFA) total scores range from 0 to 20, with higher scores reflecting a worse clinical status or outcome. An mSOFA total score of 0 or 1 reflects resolution of organ dysfunction/failure.
  score on a scale | 5.6 (2.5) | 5.4 (2.2) | 5.5 (2.4)
Acute Physiology And Chronic Health Evaluation II (APACHE II) Score [Mean (Standard Deviation); unit: score on a scale] — The Acute Physiology and Chronic Health Evaluation (APACHE) Score is a severity of illness classification system. It is determined within 24 hours of admission of a patient to an intensive care unit (ICU): an integer score from 0 to 71 is computed based on several measurements (physiologic variables, age, chronic health status). Higher scores correspond to more severe disease and a greater risk of death.
  score on a scale | 16.4 (6.8) | 16.4 (6.6) | 16.4 (6.7)
Sepsis Presentation [Count of Participants; unit: Participants] — Sepsis presentation is based on mSOFA cardiovascular and respiratory sub-score components equal to 3 or 4.
  Participants
    Cardiovascular Organ Failure | 81 | 62 | 143
    Respiratory Organ Failure | 19 | 11 | 30
Acute Kidney Injury (AKI) Presentation [Count of Participants; unit: Participants] — Stages of acute kidney injury (AKI) refer to the Kidney Disease: Improving Global Outcomes (KDIGO) stages of AKI. There are 3 KDIGO stages of AKI that are based on serum creatinine or urine output. Stage 1 represents the least severity of AKI, while Stage 3 represents the greatest severity of AKI.
  Participants
    Any AKI at Screening | 87 | 103 | 190
    Stage 2 or 3 AKI at Screening | 62 | 81 | 143

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Necrotizing Infections Clinical Composite Endpoint (NICCE)
Description: NICCE was made up of the following 5 components, all of which had to be met to successfully achieve the primary outcome measure (i.e., a "responder"): (i) Alive at Day 28, (ii) ≤ 3 debridements through Day 14, (iii) No amputation performed after the first debridement, (iv) Day 14 modified Sequential Organ Failure Assessment (mSOFA) score ≤ 1, and (v) Reduction of ≥ 3 mSOFA score points between Baseline and Day 14. This analysis compared responders in the reltecimod group versus responders in the placebo group.
  Modified Sequential Organ Failure Assessment (mSOFA) total scores range from 0 to 20, with higher scores reflecting a worse clinical status or outcome. An mSOFA total score of 0 or 1 reflects resolution of organ dysfunction/failure.
Time Frame: 28 days
Population: The primary analysis population (modified intent-to-treat [mITT]) included all randomized patients who were exposed to study drug and who had a definitive diagnosis of NSTI based on surgical verification.
  A secondary analysis of the primary outcome measure utilized the United States-modified intent-to-treat (US-mITT) analysis population which consisted only of mITT patients enrolled in the United States.
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 142 | 148
Participants
  mITT Population | 69 | 59
  US-mITT Population: number analyzed (Participants) | 135 | 138
  US-mITT Population | 67 | 50
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; This analysis utilized the mITT analysis population; Test type: Superiority; p = 0.135, Chi-squared
Statistical Analysis 2: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; This analysis utilized the US-mITT analysis population; Test type: Superiority; p = 0.025, Chi-squared

2. Secondary Outcome: Number of Patients With One or More Adverse Events (AEs)
Description: Number of Patients With One or More Adverse Events (AEs). Serious Adverse Events (SAEs) are included in this outcome measure since SAEs are a subset of AEs.
Time Frame: 28 days
Population: As Treated/Safety Analysis Population: all randomized patients who were exposed to study drug (active or placebo) and categorized according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Groups:
- AB103 0.5 mg/kg: AB103 0.5 mg/kg, IV infusion, single dose
- Placebo: NaCl 0.9%, IV infusion, single dose
Arm/Group | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 143 | 147
Participants | 104 | 96

3. Secondary Outcome: Number of Patients With One or More Serious Adverse Events (SAEs)
Description: Number of Patients with One or More Serious Adverse Events (SAEs) During the Study
Time Frame: 28 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 143 | 147
Participants | 44 | 40

4. Secondary Outcome: Number of Patients With One or More Secondary Infections
Description: Number of Patients with One or More Secondary Infections During the Study
Time Frame: 28 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 143 | 147
Participants | 30 | 32

5. Secondary Outcome: Number of Patients Achieving Day 14 Modified Sequential Organ Failure Assessment (mSOFA) Score of 0 or 1
Description: Modified Sequential Organ Failure Assessment (mSOFA) total scores range from 0 to 20, with higher scores reflecting a worse clinical status or outcome. An mSOFA total score of 0 or 1 reflects resolution of organ dysfunction/failure.
Time Frame: 14 days
Population: The United States modified intent-to-treat (US-mITT) population included all randomized patients in the United States who were exposed to study drug and who had a definitive diagnosis of NSTI based on surgical verification. This population does not include 17 patients randomized in France.
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 135 | 138
Participants | 87 | 74
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.069, Chi-squared

6. Secondary Outcome: Intensive Care Unit (ICU)-Free Days
Description: ICU-free days refers to the number of days a patient did not spend time in the ICU through Day 28.
Time Frame: 28 days
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 135 | 138
days | 20.0 [0 to 28] | 18.0 [0 to 28]
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.401, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Ventilator-free Days
Description: Ventilator-free days refers to the number of days a patient was not on a ventilator through Day 28.
Time Frame: 28 days
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 135 | 138
days | 22.0 [0 to 28] | 21.0 [0 to 28]
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.195, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Vasopressor-free Days
Description: Vasopressor-free days refers to the number of days a patient did not receive a vasopressor through Day 28.
Time Frame: 28 days
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 135 | 138
days | 25.0 [0 to 28] | 25.0 [0 to 28]
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.596, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Hospital Days
Description: Hospital days refers to the number of days a patient spent time in the hospital.
Time Frame: 90 days or until end of follow up
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 135 | 138
days | 18.0 [1 to 103] | 19.5 [2 to 135]
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.512, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Number of Patients With a More Favorable or Less Favorable Hospital Discharge Location
Description: Number of patients with more favorable discharge location (home or rehabilitation facility) or less favorable discharge location (skilled nursing facility, another acute care facility, death, other)
Time Frame: 90 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 135 | 138
Participants
  More Favorable Discharge Location | 80 | 64
  Less Favorable Discharge Location | 55 | 74
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.033, Chi-squared

11. Other Pre Specified Outcome: Number of Deaths From Day 0 Through Day 90
Description: The number of deaths occurring from Study Day 0 through Study Day 90
Time Frame: 90 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 135 | 138
Participants | 24 | 29
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.554, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.50 to 1.46]

12. Other Pre Specified Outcome: Number of Deaths After Day 14 Through Day 90
Description: Number of deaths after Study Day 14 through Study Day 90
Time Frame: 76 days (after Day 14 through Day 90)
Population: The United States modified intent-to-treat (US-mITT) population included all randomized patients in the United States who were exposed to study drug and who had a definitive diagnosis of NSTI based on surgical verification. This population does not include 17 patients randomized in France. Data from patients in the US-mITT population alive on Day 14 (119 reltecimod patients and 124 placebo patients) were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 119 | 124
Participants | 8 | 15
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.148, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.23 to 1.26]

13. Other Pre Specified Outcome: Number of Deaths From Day 0 Through Day 90 Among Patients With a Screening mSOFA Score of at Least 5
Description: Number and percentage of patients with a Screening mSOFA score of at least 5 who were alive on Study Day 0 and subsequently died through Study Day 90.
Time Frame: 90 days
Population: The United States modified intent-to-treat (US-mITT) population included all randomized patients in the United States who were exposed to study drug and who had a definitive diagnosis of NSTI based on surgical verification. This population does not include 17 patients randomized in France. Data from patients in the US-mITT population with a Screening mSOFA score of at least 5 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 77 | 79
Participants | 16 | 19
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.736, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.46 to 1.73]

14. Other Pre Specified Outcome: Number of Deaths After Day 14 Through Day 90 Among Patients With a Screening mSOFA Score of at Least 5
Description: Number and percentage of patients with a Screening mSOFA score of at least 5 who were alive on Study Day 14 and subsequently died through Study Day 90.
Time Frame: 76 days (after Day 14 through Day 90)
Population: The United States modified intent-to-treat (US-mITT) population included all randomized patients in the United States who were exposed to study drug and who had a definitive diagnosis of NSTI based on surgical verification. This population does not include 17 patients randomized in France. Data from patients in the US-mITT population with a Screening mSOFA score of at least 5 who were alive on Day 14 (64 reltecimod patients and 69 placebo patients) were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 64 | 69
Participants | 3 | 9
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.093, Log Rank; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.09 to 1.25]

15. Other Pre Specified Outcome: Number of Deaths From Day 0 Through Day 90 Among Patients With Baseline Cardiovascular Failure (Shock)
Description: Number and percentage of patients with baseline cardiovascular failure (shock) who died through Study Day 90.
Time Frame: 90 days
Population: The United States modified intent-to-treat (US-mITT) population included all randomized patients in the United States who were exposed to study drug and who had a definitive diagnosis of NSTI based on surgical verification. This population does not include 17 patients randomized in France. Data from patients in the US-mITT population with baseline cardiovascular failure (i.e., shock; 75 reltecimod patients and 56 placebo patients) were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 75 | 56
Participants | 14 | 15
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.352, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.35 to 1.46]

16. Other Pre Specified Outcome: Number of Deaths After Day 14 Through Day 90 Among Patients With Baseline Cardiovascular Failure (Shock)
Description: Number and percentage of patients with baseline cardiovascular failure (shock) who were alive on Study Day 14 and subsequently died through Study Day 90.
Time Frame: 76 days (after Day 14 through Day 90)
Population: The United States modified intent-to-treat (US-mITT) population included all randomized patients in the United States who were exposed to study drug and who had a definitive diagnosis of NSTI based on surgical verification. This population does not include 17 patients randomized in France. Data from patients in the US-mITT population with baseline cardiovascular failure (i.e., shock; 63 reltecimod patients and 48 placebo patients) were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 63 | 48
Participants | 2 | 7
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.031, Log Rank; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.04 to 0.99]

17. Other Pre Specified Outcome: Number of Patients With a Screening Modified Sequential Organ Failure Assessment (mSOFA) Score of at Least 5 Who Achieved NICCE
Description: NICCE was made up of the following 5 components, all of which had to be met to successfully achieve the primary outcome measure: (i) Alive at Day 28, (ii) ≤ 3 debridements through Day 14, (iii) No amputation performed after the first debridement, (iv) Day 14 modified Sequential Organ Failure Assessment (mSOFA) score ≤ 1, and (v) Reduction of ≥ 3 mSOFA score points between Baseline and Day 14.
  Modified Sequential Organ Failure Assessment (mSOFA) total scores range from 0 to 20, with higher scores reflecting a worse clinical status or outcome. An mSOFA total score of 0 or 1 reflects resolution of organ dysfunction/failure.
Time Frame: 28 days
Population: The United States modified intent-to-treat (US-mITT) population included all randomized patients in the United States who were exposed to study drug and who had a definitive diagnosis of NSTI based on surgical verification. This population does not include 17 patients randomized in France. Data from patients in the US-mITT population with a Screening mSOFA score of at least 5 (77 reltecimod patients and 79 placebo patients) were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 77 | 79
Participants | 38 | 25
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.024, Chi-squared

18. Other Pre Specified Outcome: Number of Patients With a Screening mSOFA Score of at Least 5 Who Achieved Day 14 Modified Sequential Organ Failure Assessment (mSOFA) Score of 0 or 1
Description: as for outcome 5
Time Frame: 14 days
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 77 | 79
Participants | 45 | 29
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.007, Chi-squared

19. Other Pre Specified Outcome: Number of Patients With Baseline Cardiovascular Failure (Shock) Who Achieved NICCE
Description: NICCE was made up of the following 5 components, all of which had to be met to successfully achieve the primary outcome measure: (i) Alive at Day 28, (ii) ≤ 3 debridements through Day 14, (iii) No amputation performed after the first debridement, (iv) Day 14 modified Sequential Organ Failure Assessment (mSOFA) score ≤ 1, and (v) Reduction of ≥ 3 mSOFA score points between Baseline and Day 14.
Time Frame: 28 days
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 75 | 56
Participants | 38 | 18
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.034, Chi-squared

20. Other Pre Specified Outcome: Number of Patients With Baseline Cardiovascular Failure (Shock) Who Achieved Day 14 Modified Sequential Organ Failure Assessment (mSOFA) Score of 0 or 1
Description: as for outcome 5
Time Frame: 14 days
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
Number analyzed (Participants) | 75 | 56
Participants | 48 | 21
Statistical Analysis 1: Comparison: Reltecimod (AB103) 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.003, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from study drug administration through the Day 28 visit. Data associated with deaths and study drug-related serious adverse events (SAEs) were collected from study drug administration though the Day 90 visit.
Description: Safety data obtained during study visits associated with Study Days 1, 2, 3, 7, 10, 14, 21, and 28 were systematically assessed throughout the study. In addition, data from spontaneously reported AEs were included in safety assessments. Data associated with deaths and study drug-related serious adverse events (SAEs) were collected from study drug administration though the Day 90 visit.
Groups:
- Reltecimod (AB103) 0.5 mg/kg: Reltecimod (AB103) 0.5 mg/kg, single IV infusion over approximately 10 minutes
Arm/Group | Reltecimod (AB103) 0.5 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 24/143 | 29/147
Serious Adverse Events (participants affected / at risk) | 44/143 | 40/147
Other Adverse Events (participants affected / at risk) | 24/143 | 25/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reltecimod (AB103) 0.5 mg/kg (N=143) | Placebo (N=147)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac arrest (Cardiac disorders) | 4 (4) | 4 (4)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 3 (3) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Organ failure (General disorders) | 2 (2) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Funguria (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Necrotizing fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Necrotizing soft tissue infection (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 2 (2)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglycemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 2 (2)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Skin discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leg amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reltecimod (AB103) 0.5 mg/kg (N=143) | Placebo (N=147)
Anemia (Blood and lymphatic system disorders) | 8 (10) | 6 (7)
Atrial fibrillation (Cardiac disorders) | 7 (7) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 8 (8)
Pneumonia (Infections and infestations) | 5 (5) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT02469857/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT02469857/SAP_001.pdf